CLINICAL TRIAL: NCT02693158
Title: Direct Implantation of Sirolimus-Eluting Stents With Bioresorbable Drug Carrier Technology Utilizing the Svelte Drug-Eluting Coronary Stent: The Direct III Post Market Study
Brief Title: The Direct III Post Market Study
Acronym: Direct III
Status: Completed | Type: Observational
Sponsor: Svelte Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IP-15-002
Record Dates: First submitted 2016-02-18; First posted 2016-02-26 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this multicenter, single-arm, observational study is to evaluate the feasibility of a systematic direct stenting strategy with the Svelte SLENDER IDS Sirolimus-Eluting Coronary Stent-on-a-Wire Integrated Delivery System (SLENDER IDS) in an all-comers, real-world population.

DETAILED DESCRIPTION:
In this post-market study, the population will include real-world subjects who are intended to be treated, with SLENDER IDS as standard therapy. Follow-up contacts post procedure will be made for clinical assessments at hospital discharge, 1, 6 and 12 months.

This study is designed as a prospective, multi-center, single-arm, observational all-comers clinical study to collect ongoing safety and efficacy of SLENDER IDS and to determine the feasibility of a direct stenting strategy in an all-comers population. A minimum of two hundred fifty (250) subjects will be treated at up to 20 sites in Europe.

Review of safety data and risks to subjects will be monitored by an independent Clinical Events Committee (CEC) at pre-specified enrollment milestones.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old;
2. Subject has symptomatic heart disease due to coronary artery lesions of length < 28 mm and a reference vessel diameter 2.5 - 4.0 mm.
3. Subject is intended to be treated with PCI and implantation of SLENDER IDS as part of his/her standard treatment
4. Subject or subject's legal representative understands the study requirements and the treatment procedures and provides written informed consent before any study specific tests or procedures are performed.

Exclusion Criteria:

1. Subject is unable to receive anti-platelet and/or anti-coagulant therapy;
2. Subject is allergic to sirolimus, PEA III Ac Bz, cobalt, chromium, nickel or tungsten;
3. The subject is judged to have lesions preventing complete inflation of an angioplasty balloon or proper placement of a coronary stent, including chronic total occlusions.
4. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential, based on the standard of care for the cath lab);
5. Subject is participating in another investigational drug or device clinical trial that the investigator feels would interfere with the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed as a prospective, multi-center, single-arm, observational all-comers clinical study to collect ongoing safety and efficacy of SLENDER IDS and to determine the feasibility of a direct stenting strategy in an all-comers population.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Cardiac Death, Target Vessel Myocardial Infarction (TVMI) (Q wave and non-Q wave) or clinically driven Target Lesion Revascularization (TLR) by percutaneous or surgical methods.

SECONDARY OUTCOMES:
Target Vessel Failure (TVF) | Discharge, 1, 6 and 12 months
  composite endpoint of Cardiac Death, Target Vessel MI, or clinically-driven Target Vessel Revascularization (TVR) by percutaneous or surgical methods.
Major Adverse Cardiac Event (MACE) | Discharge, 1, 6 and 12 months
  defined as a composite of all deaths, Target Vessel MI (Q wave and non-Q wave), emergent coronary artery bypass grafting surgery (CABG), or clinically-driven repeat Target Lesion Revascularization (TLR) by percutaneous or surgical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Donohoe, MD, Study Director — Svelte Medical
Locations (8):
- Netherlands (8):
  - Meander Medical Center, Amersfoort
  - OLVG, Amsterdam
  - Tergooi Hospital, Blaricum
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - St Antonius Hospital, Nieuwegein
  - HagaZiekenhuis, The Hague
  - University Medical Center, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided